CLINICAL TRIAL: NCT02476357
Title: A Randomized Control Trial for Lymphocele and Lymphorrhea Control Following Inguinal and Axillary Radical Lymph Node Dissection
Brief Title: A Study for Lymphocele and Lymphorrhea Control Following Inguinal and Axillary Radical Lymph Node Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, Professor, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYMPH-01
Record Dates: First submitted 2015-02-20; First posted 2015-06-19 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Lymph Node Dissection; Lymphoedema; Lymphocoele
MeSH Terms: conditions — Lymphedema; Lymphocele

STUDY DESIGN:
Intervention Model Description: Monocentric, open, interventional, randomized with two arms 1:1
Who Masked: Participant
Masking Description: unblinded
Oversight: Data Monitoring Committee: No

ARMS (2):
- Harmonic (Active Comparator): Harmonic Scalpel (HS; Ethicon Endo-Surgery, Cincinnati, OH)
  Interventions: Device: Harmonic scalpel
- Control (Active Comparator): Monopolar scalpel and ligature
  Interventions: Device: Harmonic scalpel

INTERVENTIONS:
Device: Harmonic scalpel

SUMMARY:
Patients undergoing groin or axillary Radical lymph node dissection (RLND) or completion lymph node dissection (CLND, after positive sentinel lymph node biopsy (SLNB) for melanoma or breast cancer were randomized in a controlled trial for surgical dissection technique. Harmonic scalpel dissection were compared with classic dissection in term of lymphocoele and oedema.

DETAILED DESCRIPTION:
The aim of the present study was to assess the value of USS in RLND in groin and axilla in a homogenous group of patients.

In a tertiary academic centre, patients undergoing groin or axillary RLND or CLND after positive SLNB for melanoma, skin cancer, sarcoma or breast cancer were enrolled in a randomized controlled trial for surgical dissection technique. The study was reviewed and accepted by the local ethical committee. Patients were older than 18 years and gave an informed consent. All patients with a past medical history of contralateral lymph node dissection or other cause of lymphedema (previous trauma, deep venous thrombosis, radiotherapy, etc.) were excluded. Patients undergoing both iliac and inguinal lymph node dissections were excluded as well. No patients had distant or in transit metastasis. Patients were randomly assigned using sealed numbered envelopes to one of two arms of the study in a 1: 1 ratio. In the first group the dissection was conducted with USS (Harmonic Focus ®, Ethicon Endo-Surgery (Europe) GmbH) exclusively. In the control group the lymphadenectomy was performed using ligation and monopolar electrocautery. All patients were operated by a dedicated team headed by a single surgeon.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing groin or axillary Radical lymph node dissection (RLND) or completion lymph node dissection (CLND), after positive sentinel lymph node biopsy (SLNB) for melanoma or breast cancer were included.

Exclusion Criteria:

* Patient with a past medical history of contralateral lymph node dissection or other cause for lymphedema (trauma, deep venous thrombosis, radiotherapy, etc.) were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Matter, Prof, Study Director — University of Lausanne Hospitals
Locations (1):
- Department of Visceral Surgery, University Hospital Center, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Gie O, Matthey-Gie ML, Marques-Vidal PM, Demartines N, Matter M. Impact of the Ultrasonic scalpel on the amount of drained lymph after axillary or inguinal lymphadenectomy. BMC Surg. 2017 Mar 21;17(1):27. doi: 10.1186/s12893-017-0222-1. PMID 28327108

RESULTS

PARTICIPANT FLOW:
Groups:
- Harmonic: Harmonic Scalpel (HS; Ethicon Endo-Surgery, Cincinnati, OH)
  Harmonic scalpel
- Control: Monopolar scalpel and ligature
  Harmonic scalpel
Period: Overall Study
Arm/Group | Harmonic | Control
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Harmonic | Control | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (15.1) | 61.9 (13.3) | 60.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 16 | 16 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Draining Time
Description: Duration (days) between surgery and removal of postoperative suction drain
Time Frame: Lymph quantity measured every day. Drained removed when < 50 ml. per day for 2 consecutive days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Harmonic | Control
Number analyzed (Participants) | 40 | 40
days | 31 (20) | 32 (18)

2. Secondary Outcome: Daily Amount of Drained Lymph
Description: Patients had to record on a list the amount in ml. of lymph in the suction drain bottles
Time Frame: Lymph quantity measured every day, up to 50 days.
Population: One patient in the Harmonic group was excluded due to insufficient data collection of lymph at home
Measure: Mean (Standard Deviation); unit: ml.
Arm/Group | Harmonic | Control
Number analyzed (Participants) | 39 | 40
ml. | 2908 (2453) | 3898 (5791)

ADVERSE EVENTS:
Arm/Group | Harmonic | Control
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No